CLINICAL TRIAL: NCT06701500
Title: SFB TRR 265: Losing and Regaining Control Over Drug Intake Project B03: Role of Pavlovian Mechanisms for Control Over Substance Use Project B09: Maladaptive Context Inference As Key Mechanism Underlying Impaired Control
Brief Title: Assessing Habitual, Goal-Directed, and Pavlovian Influences in Alcohol Use Disorder
Acronym: ReCoDe
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Charite University, Berlin, Germany (Other); Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Other Study IDs: 40217046123
Record Dates: First submitted 2024-09-25; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Use Disorder (AUD); Alcoholism; Substance Use Disorders
Keywords: Substance use disorder (SUD); Alcohol use disorder (AUD); Outcome-specific Pavlovian to instrumental transfer; Humans; Surveys and Questionnaires; Reward; Cues; Habit formation; Goal-directed behavior
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Alcohol Use Disorder (AUD) Group: Participants with alcohol use disorder (moderate to severe if no withdrawal symptoms)
  Interventions: Behavioral: Pavlovian-to-instrumental transfer (PIT) paradigm; Behavioral: Action Sequence Task (AST); Diagnostic Test: Basic psychological assessment (interview); Diagnostic Test: Basic psychological assessment (questionnaires); Behavioral: Neuropsychology tests
- Control Group: Participants without SUD
  Interventions: Behavioral: Pavlovian-to-instrumental transfer (PIT) paradigm; Behavioral: Action Sequence Task (AST); Diagnostic Test: Basic psychological assessment (interview); Diagnostic Test: Basic psychological assessment (questionnaires); Behavioral: Neuropsychology tests

INTERVENTIONS:
Behavioral: Pavlovian-to-instrumental transfer (PIT) paradigm — The paradigm consists of four parts:
  In the first part, an instrumental learning task is completed in which subjects must learn which stimuli require a response and which do not. In the second part, a classical (Pavlovian) conditioning task is then completed in which subjects learn by passive viewing which stimuli are associated with certain amounts of money. The third part measures to which instrumental responses (learned in Part 1) are modulated by the presentation of the classically conditioned stimuli (learned in Part 2). At the same time drug-associated stimuli are presented in the background measuring to which extent they conflict with the learned instrumental behavior. In the last part, query trials are implemented in which the participants have to choose between two pictures to assess the relative cue value.
Behavioral: Action Sequence Task (AST) — Participants need to press four keys according to the cue location; two keys are associated with high reward, while the other two are associated with low reward in case of correct and timely responses. The explicit goal is to maximize the reward. While in half of the trials the cues are presented in a random order, in the other half of the trials, participants repeatedly perform a fixed action sequence of 12 elements (habit condition). The degree of action sequence chunking (i.e. automation) is assessed via the differences in error rates and reaction times between the random and fixed order condition (habit parameter). Importantly, 15% of all trials are dual- target trials. In these the goal-directed system (press high reward key) and the action sequence (press sequence key) can either be in line (congruent trials) or in conflict (incongruent trials) with each other, thus the interference between goal-directed and habitual control can be tested.
Diagnostic Test: Basic psychological assessment (interview) — * Structured Clinical Interview for DSM Disorders (SCID) Current Depression:
    * SCID Mania
    * SCID alcohol use disorder (AUD)
    * SCID tobacco use disorder (TUD)
  * Alcohol, Smoking and Substance Involvement Screening Test (ASSIST)
  * Alcohol quantity-frequency
  * Tobacco quantity-frequency
  * Cannabis and other substances quantity-frequency
Diagnostic Test: Basic psychological assessment (questionnaires) — * Sociodemographics
  * Edinburgh Handedness Inventory (EHI)
  * Fagerström Test for Nicotine depend (FTND)
  * Barratt Impulsiveness Scale - Kurzversion (BIS-15)
  * Alcohol Use Disorders Identification Test (AUDIT)
  * Cannabis Use Disorders Identification Test (CUDIT)
  * Adult ADHD Self-Report Scale (ASRS)
Behavioral: Neuropsychology tests — * Digit-Symbol-Test (DST)
  * Go/Nogo Simon task
  * Counting Stroop Task
  * Value-based decision-making task (VBDM)

SUMMARY:
The first aim of this study is to establish the role of maladaptive reliance on habits for impaired control in addiction, employing a novel task - the Action-Sequence-Task (AST), which assesses interference between habitual and goal-directed control. The AST, along with the developed computational model, will be employed to test whether participants with Alcohol Use Disorder (AUD) and control participants differ with respect to task performance and estimated model parameters. The investigators hypothesize stronger habitual behavior (increased habitual tendency) and an increased susceptibility to conflict between habitual and goal-directed control, measured as increased interference, are associated with AUD.

The second aim of the study is to understand whether Pavlovian-to-Instrumental Transfer (PIT) reflects more of a controlled, goal-directed process, or a more automatic, habitual process. The investigators will use the single-lever PIT task as it is an efficient tool for testing the interaction between Pavlovian cues and instrumental behavior, especially when they are in conflict. In these trials, top-down control must be allocated to successfully overcome the conflict, which may share some common underlying mechanisms with the arbitration between goal-directed and habitual behavior during conflict, as assessed by the novel AST. The third aim of the study is to investigate whether severely dependent AUD patients would show a stronger PIT effect compared to a control group, consistent with the investigators' previous findings.

DETAILED DESCRIPTION:
This project has three research aims:

1. Investigate whether stronger habitual behavior and increased susceptibility to the conflict between habitual and goal-directed control are associated with SUD
2. Investigate whether PIT is more of a habitual or a goal-directed process.
3. Replicate the previous findings that moderate to severely dependent AUD patients show a stronger PIT effect in contrast to the control group The experiment will be conducted in 90 AUD patients and 90 age and gender-matched controls. Participants will perform the AST task over two consecutive days, and during the second day, they will also perform the single-lever PIT task. In the AST, participants need to press four keys according to the cue location; two keys are associated with high reward, while the other two are associated with low reward in case of correct and timely responses. The explicit goal is to maximize the reward. While in half of the trials the cues are presented in a random order, in the other half of the trials, participants repeatedly perform a fixed action sequence of 12 elements (habit condition). The degree of action sequence chunking (i.e. automation) is assessed via the differences in error rates and reaction times between the random and fixed order condition (habit parameter). Importantly, 15% of all trials are dual- target trials. In these, the goal-directed system (press high reward key) and the action sequence (press sequence key) can either be in line (congruent trials) or in conflict (incongruent trials) with each other. Thus, the interference between goal-directed and habitual control can be tested.

The single-lever PIT task consists of four phases. In the instrumental task, participants need to learn which shells to collect or leave in order to gain as much money as possible; the correct choice is probabilistically rewarded in 80% of all times. During the Pavlovian conditioning phase, colorful fractals are presented in the back of the screen, which have been passively paired either with monetary loss, no change or monetary gain, i.e. they act as positively valued, neutral or negatively valued cues. During the transfer phase, participants were instructed to perform the instrumental task as they have done previously. These fractals thus act as independent, Pavlovian conditioned background stimuli and interact with instrumental behavior in the unrelated task to collect the correct shells. To avoid further learning, this transfer part will be conducted under nominal extinction. Finally, query trials, in which one of two pictures will have to be chosen, will be used to assess the relative cue value.

The participants will additionally perform a Counting Stroop task and a No-go Simon task. In the Stroop task, either one, two, three or four identical digits from 1 to 4 are shown. Number and denotation of digits are either congruent (1, 22, 333, 4444; 80 trials) or incongruent (111, 2222, 3, 44; 80 trials). Subjects have to indicate how many digits were shown. In the No-go Simon task, the investigators will show arrows either pointing to the left or right. The arrow can either be shown on the left or the right side of the display. In congruent trials, direction and position are the same, whereas they differ in incongruent trials. Participants have to indicate the direction of the arrow and ignore the position. 20% of trials are No-go trials, indicated by bold arrows. Here subjects have to always withhold a response (inhibition task).

Expected results:

Hypothesis a: The investigators hypothesize an increased habitual tendency and susceptibility to conflict, i.e. interference between habitual and goal-directed control as assessed with the AST in AUD participants. More specifically, the investigators hypothesize that the AUD participants will perform the fixed sequence faster and with fewer errors on the second day of AST. Moreover, in contrast to the control group, AUD participants will choose the high reward keys less often in incongruent trials (when the goals-directed control and the habitual action sequence are in conflict with each other), indicating a shift from goal-directed to habitual control.

Hypothesis b: Given that the allocation of top-down control is needed for overcoming interference by Pavlovian cues and exhibiting more goal-directed control, the investigators expect that participants with stronger PIT effect (lower interference control) also acquire habits more easily and show increased habitual control. Additionally, the investigators hypothesize that the participants with a higher PIT effect will exhibit a shift from goal-directed to habitual control, as indicated by a lower frequency of high reward keys in incongruent trials. As a general process, these associations should be observable in both, the AUD and the control group.

Hypothesis c: As a replication, the investigators expect the AUD group to show a stronger PIT effect in contrast to the control group.

Hypothesis d: Both Interference costs (i.e. increased ER in instrumental responses) during PIT and interference costs between goal-directed and habitual behavior will be associated with interference costs at the stimulus level (Stroop task) and at the response level (No-go Simon task), and these costs will also be correlated with the ER during response inhibition (No-go Simon task).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* AUD subjects only: meet 4 or more criteria for DSM-5 alcohol use disorder
* Sufficient motor skills and visual acuity to use PC
* Ability to consent to the study and complete the questionnaires
* Sufficient German skills

Exclusion Criteria:

* Lifetime diagnosis of DSM-5 bipolar disorder, schizophrenia or schizophrenia spectrum disorder
* Current diagnosis of severe major depression according to DSM-5, or presence of suicidal intention
* Pregnancy
* Severe withdrawal symptoms
* Acute drug intoxication at the appointments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants recruited through the addiction in- and outpatient clinic of University Hospital Dresden as well as from our partner clinic in Radebeul.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-03-02 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Behavioral single-lever Pavlovian to instrumental transfer (PIT) effect | 1 day, 1 hour
  Strength of interference PIT effect assessed with the single-lever PIT paradigm: increased error rate in the incongruent condition as compared with the congruent condition.
Action Sequence Task (AST) day one and day two | 2 days, 1 hour per day
  Habit formation: faster response time and decreased errors of preforming fixed compared to the random action sequence. Shift from goal-directed to habitual control: less choices of the high reward keys in trials in the incongruent trials where the goal-directed control and the habitual action sequence are in conflict (incongruent trials)

SECONDARY OUTCOMES:
Counting Stroop task | 1 day, 10 minutes
  Interference cost at the stimulus level: increased error rate in the incongruent condition as compared with the congruent condition.
Go-Nogo Simon task | 1 day, 20 minutes
  Interference cost at the response level: increased error rate in the incongruent condition as compared with the congruent condition. Response inhibition: error rate during No-go trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Technische Universität Dresden, Dresden, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Belanger MJ, Chen H, Hentschel A, Garbusow M, Ebrahimi C, Knorr FG, Zech HG, Pilhatsch M, Heinz A, Smolka MN. Development of Novel Tasks to Assess Outcome-Specific and General Pavlovian-to-Instrumental Transfer in Humans. Neuropsychobiology. 2022;81(5):370-386. doi: 10.1159/000526774. Epub 2022 Nov 14. PMID 36380640
- [Background] Frolich S, Esmeyer M, Endrass T, Smolka MN, Kiebel SJ. Interaction between habits as action sequences and goal-directed behavior under time pressure. Front Neurosci. 2023 Jan 13;16:996957. doi: 10.3389/fnins.2022.996957. eCollection 2022. PMID 36711151
- [Background] Kronke KM, Wolff M, Benz A, Goschke T. Successful smoking cessation is associated with prefrontal cortical function during a Stroop task: A preliminary study. Psychiatry Res. 2015 Oct 30;234(1):52-6. doi: 10.1016/j.pscychresns.2015.08.005. Epub 2015 Aug 20. PMID 26321462
- [Background] Chmielewski WX, Beste C. Testing interactive effects of automatic and conflict control processes during response inhibition - A system neurophysiological study. Neuroimage. 2017 Feb 1;146:1149-1156. doi: 10.1016/j.neuroimage.2016.10.015. Epub 2016 Oct 11. PMID 27742599